CLINICAL TRIAL: NCT01161537
Title: A Phase 2, Single-Blind, Placebo-Controlled Study to Evaluate the Effect of VX-770 on Hyperpolarized Helium-3 Magnetic Resonance Imaging in Subjects With Cystic Fibrosis, the G551D Mutation, and FEV1 ≥40% Predicted
Brief Title: Study of the Effect of VX-770 on Hyperpolarized Helium-3 Magnetic Resonance Imaging in Subjects With Cystic Fibrosis and the G551D Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VX10-770-107
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Results first posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VX-770 (Experimental): Part A: Subjects received placebo tablets matched to VX-770 150 milligram (mg) orally twice daily from Day 1 to 14 (Placebo run-in period), followed by VX-770 150 mg tablets orally twice daily from Day 15 to 42 (VX-770 treatment period), and then placebo tablets matched to VX-770 150 mg orally twice daily from Day 43 to 57 (Placebo washout period) during Part A of the study.
  Part B: Subjects received VX-770 150 mg tablets orally twice daily for 48 weeks during Part B of the study. Part B included subjects from Part A and newly enrolled subjects.
  Interventions: Drug: VX-770; Drug: Placebo

INTERVENTIONS:
Drug: VX-770 — Tablet.
  Other Names: Ivacaftor
Drug: Placebo — Tablet.

SUMMARY:
Cystic Fibrosis (CF) is caused by mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene. The encoded protein, CFTR, is an epithelial chloride ion channel responsible for aiding in the regulation of salt and water absorption and secretion in various tissues. Although the disease affects multiple organs, the leading cause of mortality is the progressive loss of lung function. Obstruction of airways with thick mucus, chronic bacterial infection of the airways, and inflammatory response are all thought to play a role in causing lung damage. Through its function as a chloride channel, CFTR is believed to be integral in epithelial ion and water transport and hence, maintaining the normal hydration of lung secretions.

VX-770 (ivacaftor) is a potent and selective potentiator of wild-type, G551D, F508del, and R117H forms of human CFTR. Based on in vitro studies and pharmacologic, pharmacokinetic (PK), and safety profiles, VX-770 has been selected for clinical development as a possible treatment for patients with CF.

Hyperpolarized noble gas magnetic resonance imaging (HG-MRI) is a promising new means of assessing lung function by direct imaging of certain non-radioactive isotopes of an inert noble gas, such as helium or xenon. Through this technique, high-resolution 3-dimensional images of lung ventilation can be obtained in both pediatric and adult patients during a single short breath-hold following inhalation of the gas.

This is a 2-part study to evaluate the effect of VX-770 on hyperpolarized helium-3 magnetic resonance imaging (3He-MRI), and to evaluate the safety and efficacy of VX-770 in subjects aged 12 years and older with CF who have the G551D-CFTR mutation. Part A is a single-blind, placebo-controlled study that includes 4 weeks of VX-770 treatment and 4 weeks of placebo treatment. Part B is an open-label, 48 week study of long-term effect of VX 770 on hyperpolarized 3He-MRI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with Cystic Fibrosis
* Must have the G551D-CFTR mutation on at least 1 allele
* FEV1 ≥40% of predicted normal for age, gender, and height at Screening
* 12 years of age or older
* Must be able to swallow tablets

Exclusion Criteria:

* History of solid organ or hematological transplantation
* Ongoing participation in another therapeutic clinical study or prior participation in an investigational drug study within the 30 days prior to screening
* Use of inhaled hypertonic saline treatment within 14 days prior to the Screening Visit
* Extensive body tattoos or other physical features that will confound MRI

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Talissa Altes, MD, Principal Investigator — University of Virginia
Locations (1):
- Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Altes TA, Johnson M, Fidler M, Botfield M, Tustison NJ, Leiva-Salinas C, de Lange EE, Froh D, Mugler JP 3rd. Use of hyperpolarized helium-3 MRI to assess response to ivacaftor treatment in patients with cystic fibrosis. J Cyst Fibros. 2017 Mar;16(2):267-274. doi: 10.1016/j.jcf.2016.12.004. Epub 2017 Jan 26. PMID 28132845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was initiated on October 10, 2010 after first eligible subject signed informed consent form and enrolled in study.
Pre-assignment Details: All results were planned to be reported separately for Part A and Part B of the study.
Period: Part A
Arm/Group | VX-770
Started | 8
Completed | 8
Not Completed | 0
Period: Part B
Arm/Group | VX-770
Started | 9 (4 subjects from Part A continued in Part B of the study.)
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) = all enrolled subjects who received at least 1 dose of study drug (VX-770 or placebo in Part A and VX-770 in Part B).
Groups:
- VX-770: Part A: Subjects received placebo tablets matched to VX-770 150 mg orally twice daily from Day 1 to 14 (Placebo run-in period), followed by VX-770 150 mg tablets orally twice daily from Day 15 to 42 (VX-770 treatment period), and then placebo tablets matched to VX-770 150 mg orally twice daily from Day 43 to 57 (Placebo washout period) during Part A of the study.
  Part B: Subjects received VX-770 150 mg tablets orally twice daily for 48 weeks during Part B of the study. Part B included subjects from Part A and newly enrolled subjects.
Arm/Group | VX-770
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] — Data was planned to be reported separately for Part A and Part B of the study. Here "n" signifies participants who were evaluable for specified part of the study.
  years
    Part A (n = 8) | 18.9 (4.64)
    Part B (n = 9) | 24.4 (10.3)
Sex/Gender, Customized [Number; unit: participants] — Data was planned to be reported separately for Part A and Part B of the study. Here "n" signifies subjects who were evaluable for specified part of the study. Subjects may be counted in more than one category.
  participants
    Part A: Female (n = 8) | 4
    Part A: Male (n = 8) | 4
    Part B: Female (n = 9) | 3
    Part B: Male (n = 9) | 6
Race/Ethnicity, Customized [Number; unit: participants] — Data was planned to be reported separately for Part A and Part B of the study. Here "n" signifies subjects who were evaluable for specified part of the study. Subject may be counted in more than one category.
  participants
    Part A, Race: White (n = 8) | 7
    Part A, Race: Black or African American (n = 8) | 1
    Part A, Ethnicity: Not Hispanic or Latino (n = 8) | 8
    Part B, Race: White (n = 9) | 9
    Part B, Ethnicity: Not Hispanic or Latino (n = 9) | 9
Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) [Number; unit: participants] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Predicted FEV1 (for age, gender, and height) was calculated using the Knudson method. Number of subjects in each percent predicted FEV1 category (less than [<] 70%, greater than or equal to [>=] 70%-<90%, and >=90%) are reported. Data was planned to be reported separately for Part A and Part B of the study. Here "n" signifies subjects who were evaluable for specified part of the study. Subjects may be reported in more than one category.
  participants
    Part A: <70% (n = 8) | 2
    Part A: >=70%-<90% (n = 8) | 1
    Part A: >=90% (n = 8) | 5
    Part B: <70% (n = 9) | 6
    Part B: >=70%-<90% (n = 9) | 1
    Part B: >=90% (n = 9) | 2
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Data was planned to be reported separately for Part A and Part B of the study. Here "n" signifies subjects who were evaluable for specified part of the study.
  kilogram (kg)
    Part A (n = 8) | 66.31 (14.393)
    Part B (n = 9) | 66.53 (13.693)
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Data was planned to be reported separately for Part A and Part B of the study. Here "n" signifies subjects who were evaluable for specified part of the study.
  centimeter (cm)
    Part A (n = 8) | 167.5 (9.66)
    Part B (n = 9) | 169.9 (11.82)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI = (Weight [in kg]) divided by (Height [in meters])^2. Data was planned to be reported separately for Part A and Part B of the study. Here "n" signifies subjects who were evaluable for specified part of the study.
  kilogram per square meter (kg/m^2)
    Part A (n = 8) | 23.44 (3.570)
    Part B (n = 9) | 22.96 (4.066)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Baseline in Total Ventilation Defect Defined by Hyperpolarized Helium 3 Magnetic Resonance Imaging (3He-MRI) at Day 43
Description: Subjects inhaled hyperpolarized helium-3 (3He) gas mixed with nitrogen to make a total volume of approximately one-third forced vital capacity (FVC) to a maximum of 1 liter and hold their breath for 20 seconds or less. Rapid magnetic resonance imaging (MRI) was performed during inhalation/exhalation and/or breath-hold. Areas of decreased ventilation were observed as ventilation defects that are visualized as decreased (and/or absent) 3He intensity in 3He-MRI. The total ventilation defect was defined as the ratio of total ventilation defect volume (L) to total lung volume (L), expressed as a percentage. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug in VX-770 treatment phase (Day 15 to 42).
Time Frame: Part A: Baseline (pre-dose Day 15), Day 43
Population: FAS for Part A = all enrolled subjects who received at least 1 dose of study drug (VX-770 or placebo) in Part A.
Measure: Mean (Standard Deviation); unit: percentage of total lung volume
Arm/Group | VX-770
Number analyzed (Participants) | 8
percentage of total lung volume | -8.20 (9.013)

2. Primary Outcome: Part B: Change From Baseline in Total Ventilation Defect Defined by Hyperpolarized Helium 3 Magnetic Resonance Imaging (3He-MRI) at Week 48
Description: Subjects were asked to inhale hyperpolarized 3 He gas mixed with nitrogen to make a total volume of approximately one-third forced vital capacity (FVC) to a maximum of 1 liter and hold their breath for 20 seconds or less. Rapid MRI was performed during inhalation/exhalation and/or breath-hold. Areas of decreased ventilation were observed as ventilation defects that are visualized as decreased (and/or absent) 3He intensity in 3He MRI. The total ventilation defect was defined as the ratio of total ventilation defect volume (L) to total lung volume (L), expressed as a percentage. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug in Part B (48 weeks).
Time Frame: Part B: Baseline (Day -1), Week 48
Population: FAS for Part B = all enrolled subjects who received at least 1 dose of study drug (VX-770) in Part B.
Measure: Mean (Standard Deviation); unit: percentage of total lung volume
Arm/Group | VX-770
Number analyzed (Participants) | 9
percentage of total lung volume | -6.33 (11.859)

3. Secondary Outcome: Part A: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Related AEs
Description: AE: any adverse change from subject's baseline (pre-treatment) condition, including any adverse experience, abnormal recording/clinical laboratory assessment which occurs during course of study, whether it is considered related to study drug or not. SAE: medical event or condition, which falls into any of following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolonged hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect, important medical event.
  Related AEs includes all AEs for which the causality was either related to study drug or possibly related to study drug.
Time Frame: Part A: Day 1 up to Day 57
Population: Safety Set for Part A = all enrolled subjects who received at least 1 dose of study drug (VX-770 or placebo) in Part A. Data was reported as per the intervention received (Placebo [Placebo Run in/Washout] or VX-770 [VX-770 Treatment]).
Measure: Number; unit: participants
Groups:
- Part A Placebo Run in/Washout: Subjects who received placebo tablets matched to VX-770 150 mg orally twice daily from Day 1 to 14 (Placebo run-in period) and from Day 43 to 57 (Placebo washout period) during Part A of the study were assessed between Day 1 to 14 and Day 43 to 57 of Part A.
- Part A VX-770 Treatment: Subjects who received VX-770 150 mg tablets orally twice daily from Day 15 to 42 (VX-770 treatment period), during Part A of the study were assessed between Day 15 to 42 of Part A.
Arm/Group | Part A Placebo Run in/Washout | Part A VX-770 Treatment
Number analyzed (Participants) | 8 | 8
participants
  AEs | 2 | 3
  SAEs | 0 | 0
  Related AEs | 0 | 0

4. Secondary Outcome: Part A: Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) at Day 43
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Predicted FEV1 (for age, gender, and height) was calculated using the Knudson method. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug in VX-770 treatment phase (Day 15 to 42).
Time Frame: Part A: Baseline (pre-dose Day 15), Day 43
Population: FAS for Part A = all enrolled subjects who received at least 1 dose of study drug (VX-770 or placebo) in Part A.
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Arm/Group | VX-770
Number analyzed (Participants) | 8
percent predicted of FEV1 | 12.78 (9.203)

5. Secondary Outcome: Part A: Absolute Change From Baseline in Sweat Chloride at Day 43
Description: Sweat samples were collected using an approved Macroduct (Wescor, Logan, Utah) collection device. A volume of greater than or equal to (>=) 15 microliter was required for determination of sweat chloride. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug in VX-770 treatment phase (Day 15 to 42).
Time Frame: Part A: Baseline (pre-dose Day 15), Day 43
Population: FAS for Part A = all enrolled subjects who received at least 1 dose of study drug (VX-770 or placebo) in Part A.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | VX-770
Number analyzed (Participants) | 8
millimole per liter (mmol/L) | -42.31 (13.475)

6. Secondary Outcome: Part A: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score At Day 43
Description: The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for subjects with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug in VX-770 treatment phase (Day 15 to 42).
Time Frame: Baseline (pre-dose Day 15), Day 43
Population: FAS for Part A = all enrolled subjects who received at least 1 dose of study drug (VX-770 or placebo) in Part A.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VX-770
Number analyzed (Participants) | 8
units on a scale | -7.64 (27.529)

7. Secondary Outcome: Part B: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Related AEs
Description: as for outcome 3
Time Frame: Part B: Day 1 up to Week 48
Population: Safety Set for Part B = all enrolled subjects who received at least 1 dose of study drug (VX-770 or placebo) in Part B.
Measure: Number; unit: participants
Groups:
- Part B VX-770 Treatment: Subjects who received VX-770 150 mg tablets orally twice daily for 48 weeks during Part B of the study were assessed between Day 1 to Week 48 of Part B. Part B included subjects from Part A and newly enrolled subjects.
Arm/Group | Part B VX-770 Treatment
Number analyzed (Participants) | 9
participants
  AEs | 6
  SAEs | 1
  Related AEs | 4

8. Secondary Outcome: Part B: Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) at Week 48
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Predicted FEV1 (for age, gender, and height) was calculated using the Knudson method. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug in Part B (48 weeks).
Time Frame: Part B: Baseline (Day -1), Week 48
Population: FAS for Part B = all enrolled subjects who received at least 1 dose of study drug (VX-770) in Part B. Here, "Number of participants analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Arm/Group | VX-770
Number analyzed (Participants) | 8
percent predicted of FEV1 | 5.17 (9.422)

9. Secondary Outcome: Part B: Absolute Change From Baseline in Sweat Chloride at Week 48
Description: Sweat samples were collected using an approved Macroduct (Wescor, Logan, Utah) collection device. A volume of greater than or equal to (>=) 15 microliter was required for determination of sweat chloride. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug in Part B (48 weeks).
Time Frame: Part B: Baseline (Day -1), Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | VX-770
Number analyzed (Participants) | 8
mmol/L | -48.88 (22.271)

10. Secondary Outcome: Part B: Absolute Change From Baseline in in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score At Week 48
Description: The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for subjects with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug in Part B (48 weeks).
Time Frame: Part B: Baseline (Day -1), Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VX-770
Number analyzed (Participants) | 7
units on a scale | 15.08 (7.667)

ADVERSE EVENTS:
Time Frame: Part A: Day 1 through Day 57; Part B: Day 1 through Week 48
Description: A Participant with multiple events within a system organ class or preferred term was counted only once within the system organ class or preferred term, respectively.
Arm/Group | Part A Placebo Run in/Washout | Part A VX-770 Treatment | Part B VX-770 Treatment
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/9
Other Adverse Events (participants affected / at risk) | 2/8 | 3/8 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Placebo Run in/Washout (N=8) | Part A VX-770 Treatment (N=8) | Part B VX-770 Treatment (N=9)
INFECTIVE PULMONARY EXACERBATION OF CYSTIC FIBROSIS (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Placebo Run in/Washout (N=8) | Part A VX-770 Treatment (N=8) | Part B VX-770 Treatment (N=9)
CYSTIC FIBROSIS LUNG (Congenital, familial and genetic disorders) | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1
PAIN (General disorders) | 1 | 0 | 1
PYREXIA (General disorders) | 0 | 0 | 2
HEADACHE (Nervous system disorders) | 0 | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 4
INFECTIVE PULMONARY EXACERBATION OF CYSTIC FIBROSIS (Infections and infestations) | 0 | 0 | 2
BRONCHITIS (Infections and infestations) | 0 | 0 | 1
LABYRINTHITIS (Infections and infestations) | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 1
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 0 | 1
BODY MASS INDEX INCREASED (Investigations) | 0 | 0 | 2
SPIROMETRY ABNORMAL (Investigations) | 0 | 0 | 2
BACTERIAL TEST POSITIVE (Investigations) | 0 | 0 | 1
CERUMEN IMPACTION (Ear and labyrinth disorders) | 0 | 0 | 1
STRESS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.